CLINICAL TRIAL: NCT00495430
Title: Passive Acoustic Imaging With the Vibration Response Imaging Device in Healthy Subjects
Brief Title: Vibration Response Imaging in Healthy Subjects
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Deep Breeze (Industry)
Responsible Party: Merav Gat/VP Clinical Affairs, Deep Breeze
Other Study IDs: DB013
Record Dates: First submitted 2007-07-01; First posted 2007-07-03 (Estimated); Last update posted 2009-06-16 (Estimated); Status verified 2009-06

CONDITIONS: Healthy
Keywords: Healthy; Lung sounds; Breath sounds
MeSH Terms: conditions — Respiratory Sounds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary purpose is to test intersubject variability and establish the qualitative features of normal VRI images and the range of normality of the VRI quantitative lung data values that may be used to differentiate normal from abnormal breath sound distribution. Our hypothesis was that VRI breath sound images of healthy subjects are similar in a qualitative and quantitative manner.

DETAILED DESCRIPTION:
Computerized analyses have shown that normal lung sounds have distinctive characteristic that can be differentiated from abnormal lung sounds.However, technical issues and complicated display modes have restricted the use of computerized lung sound analyses in the clinical environment.

The VRI provides dynamic gray-scale images and quantitative lung data showing the breath sound distribution of healthy individuals. Typical features that are discerned by trained raters and quantitative lung data may serve as a reference for comparison to abnormal breath sound images.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to read, understands, and provides written Informed Consent;
* Male or Female in the age range of 18-85 years;
* Subject is healthy and has not exhibited symptoms of acute respiratory tract disease for the past two months;
* Subject has normal chest X-ray and normal lung function during the past 6 months that were judged stable;
* BMI > 21.

Exclusion Criteria:

* Subject has a history of a chronic condition that affects the lungs or heart (e.g.chronic obstructive pulmonary disease, asthma, congestive heart failure) or is suspected of having such a condition;
* Subject has a chest cage deformation;
* Subject has spine deformation (including severe scoliosis);
* Subject is Hirsute;
* Subject has a skin lesion (potentially contagious) on the back;
* Subject has a cardiac pacemaker or implantable defibrillator;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects who presented for complete physical examination as required by place of employment. Convenience sample - consecutive healthy subjects who meet study criteria are included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2004-12; Study Completion 2009-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mordechai Yigla, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Medical Center, Haifa, Israel

REFERENCES:
- [Background] Dellinger RP, Parrillo JE, Kushnir A, Rossi M, Kushnir I. Dynamic visualization of lung sounds with a vibration response device: a case series. Respiration. 2008;75(1):60-72. doi: 10.1159/000103558. Epub 2007 Jun 4. PMID 17551264
- [Background] Ploysongsang Y, Iyer VK, Ramamoorthy PA. Reproducibility of the vesicular breath sounds in normal subjects. Respiration. 1991;58(3-4):158-62. doi: 10.1159/000195918. PMID 1745848